CLINICAL TRIAL: NCT06884475
Title: Evaluation of Implantoplasty in the Treatment of Peri-Implantitis: Clinical, Inflammatory, Titanium Analysis in Crevicular Fluid and Microbiological Profile
Brief Title: Evaluation of Implantoplasty in the Treatment of Peri-Implantitis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Renato Casarin, Professor, supervisor responsible for research, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 83149424.7.0000.5418
Record Dates: First submitted 2025-02-18; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Peri-Implantitis and Peri-implant Mucositis
Keywords: Peri-implantitis; Implantoplasty; Titanium; Immune response; Microbiota; Surgical access
MeSH Terms: conditions — Peri-Implantitis | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Implantoplasty: treatment of peri-implantitis. (Experimental): After patient selection, 20 individuals (chosen randomly) will be selected to receive treatment for Peri-implantitis with surgical access and implantoplasty.
  Interventions: Procedure: Implantoplasty
- Surgical access: treatment of peri-implantitis. (Experimental): After patient selection, 20 individuals (chosen randomly) will be selected to receive treatment for peri-implantitis with surgical access and debridement without performing implantoplasty.
  Interventions: Procedure: Surgical access

INTERVENTIONS:
Procedure: Implantoplasty — Following clinical and radiographic examinations and thorough case planning, surgical procedures were performed under local anesthesia by a operator. After, anesthesia, surgical access will be performed for debridement and implantoplasty of the affected dental implant.
  Arms: Implantoplasty: treatment of peri-implantitis.
Procedure: Surgical access — Following clinical and radiographic examinations and thorough case planning, surgical procedures were performed under local anesthesia by a operator. After, anesthesia, only surgical access will be performed for debridement without implantoplasty of the affected dental implant.
  Arms: Surgical access: treatment of peri-implantitis.

SUMMARY:
The aim of this longitudinal study is to evaluate the clinical impact of implantoplasty in the treatment of peri-implantitis, exploring the potential effect of removing compromised implants on periodontal health and its correlation with the presence of titanium particles in the crevicular fluid. In addition, we seek to investigate changes in the peri-implant microbiological profile before and after implantoplasty, allowing a more comprehensive understanding of the effects of this procedure at both the biological and clinical levels, considering microbiological factors and the relationship with titanium, inflammation and peri-implant health. Forty participants diagnosed with peri-implantitis will be selected (n = 20 in each group) to participate in the study. They will be randomly allocated into two groups, according to the treatment to be performed (implantoplasty group and surgical access group for scaling). Using a millimeter-diameter periodontal probe, the initial clinical parameters of patients with periodontal and peri-implant disease will be evaluated. Biofilm and crevicular fluid will then be collected using sterile paper cones from one implant of each patient in all groups at follow-up intervals of 1, 3 and 6 months for subsequent processing and evaluation of the data. The integration of these analyses aims to offer valuable insights to optimize peri-implantitis treatment strategies, aiming at the health and longevity of dental implants.

DETAILED DESCRIPTION:
1. Participants: Adult patients diagnosed with peri-implantitis (Caton et al. 2018, Papapanou et al. 2018) will be included; Patients will be recruited from the population studied in the aforementioned case-control study, who were diagnosed with peri-implantitis; Inclusion and exclusion criteria will follow the criteria previously defined in the case-control study.
2. Participant Allocation: Participants will be randomly allocated into two groups: Group 1 (Implantoplasty) and Group 2 (Surgical Access). - Allocation will be performed by a computerized randomization system (sealed envelope.com).
3. Clinical Procedures: Group 1 (Implantoplasty): The affected implants will undergo implantoplasty, involving the remodeling of the implant surface to facilitate cleaning and remove compromised areas. Group 2 (Surgical Access): The affected implants will be treated through surgical access, with mechanical removal of the inflamed tissue and cleaning of the implant surface.
4. Clinical Evaluation: Initial clinical parameters will be recorded before the procedure and at specific intervals (1, 3 and 6 months after the procedure); Periodontal and peri-implant indices, including plaque index, bleeding on probing, probing depth and clinical attachment level, will be evaluated by a calibrated examiner.
5. Biofilm (Microbiome) Collection and Analysis: Periodontal and peri-implant biofilm samples will be collected for taxonomic analysis. All samples will be obtained prior to the periodontal examination. Prior to subgingival/submucosal biofilm collection, supragingival/supramucosal biofilm will be carefully removed using sterile curettes. The site will be isolated using cotton rolls and gently dried with an air syringe to avoid contamination with saliva. Biofilm samples will be obtained by standard filter paper points from the buccal surfaces of the teeth/implants. The filter paper points will be inserted into the gingival/peri-implant sulcus and left in place for 30 seconds. Paper spots will be placed in a microcentrifuge tube containing Tris-EDTA solution. All samples will be immediately frozen and stored at -20°C until laboratory analysis. Biofilm samples will be removed from the paper strips by adding 200 µL of phosphate-buffered saline (PBS) and vortexing for 1 minute. The paper spot will be removed and DNA isolated using the Qiagen MiniAmp kit (Valencia, CA) following the manufacturer's recommendations. Oral prophylaxis or nonsurgical periodontal treatment will not be initiated prior to sample collection, and subjects will be enrolled in a periodontal treatment program as needed.

   DNA Sequencing and Data Analysis: The V3-V4 hypervariable region of the 16S rRNA gene will be amplified using the primers and PCR conditions previously described by Klindworth et al. (2013). According to the manufacturer's recommendation, PCR purification will be performed using magnetic beads (AMPUre XP Bead, Beckman Agencourt) at a ratio of 0.8 beads/PCR volume. After ligation of the adapters, a new PCR purification will be performed using magnetic beads (AMPUre XP Bead, Beckman Agencourt) at a ratio of 1.12 beads/PCR volume. Library normalization will be performed using the SequalPrep™ Normalization Plate kit (96) (Applied Biosystems™), and the combined library will be quantified. Equimolar DNA concentrations will be pooled and sequenced on the Illumina Miseq platform to produce 300-bp paired-end sequences. Bioinformatic analysis will be performed using QIIME 2 2020.6 (Bolyen et al., 2019). Demultiplexed FASTQ files will be obtained from the sequencing facility, and q2 cutadapt (Martin, 2011) will be used to remove primers prior to the denoising process, which will be performed with q2-DADA2 (Callahan et al., 2016). The align-to-tree mafft-fasttree (q2-phylogeny) pipeline will be used to align all amplicon sequence variants (ASVs) with mafft (Katoh et al., 2002) and to construct a phylogeny with fasttree2 (Price et al., 2010). Taxonomy will be assigned to ASVs using the naive Bayes taxonomy classifier q2-feature-classifier (Bokulich et al. 2018a) trained against the Expanded Human Oral Microbiome Database (eHOMD, V15.2) (Escapa et al., 2018). Alpha-diversity metrics (Shannon (Spellerberg, 2003)), beta-diversity metrics (weighted UniFrac (Lozupone et al. 2007), unweighted UniFrac (Lozupone et al. 2005)), and Principal Coordinates Analysis (PCoA) will be estimated using the q2-diversity core-metrics-phylogenetic pipeline after samples are rarefied to 10591 sequences per sample. Differences in alpha diversity (differences within samples) will be measured using pairwise differences (Bokulich et al. 2018b). For beta diversity (differences between samples), differences between groups will be measured using permanova and permdisp (q2-diversity) tests. The core microbiome (considering the core microbiome as species present in at least 50% of the samples in a group) will be calculated using the core features from the q2-feature-table species-level table. Visualization will be performed using the q2-feature-table heatmap (to visualize the relative abundance of species) and PhyloToAST (Dabdoub et al., 2016). Differential abundance between species will be calculated using ANCOM-BC (Lin & Peddada, 2020).
6. Inflammatory Analysis: Peri-implant crevicular fluid and granulation tissue from debridement will be collected from all individuals involved in the study, at sites treated with peri-implantitis. During collection of the material, the site in question will be properly isolated and dried with sterilized cotton rolls. The supragingival biofilm will be removed and samples of gingival fluid will be obtained by inserting paper points between the tooth and the periodontal tissue interface for 30 seconds (Casarin et al. 2010). Two paper points will be used per site to obtain an adequate volume of crevicular fluid. The volume of collected fluid will be measured with the Periotron (Periotron 8000, Proflow Inc., Amityville, NY, USA) and the paper spots will then be placed in microcentrifuge tubes (Eppendorf), coded for each individual and experimental periods with 150 µL of phosphate buffer solution (PBS) and 0.05% Tween-20. The granulation tissue removed during implant scraping will be stored in RNAlater and frozen at -80C. The samples will be stored for later analysis. Before analysis, the samples will be diluted in 60 µL of buffer from the Millipore kit, vortexed for 30 minutes and then centrifuged for 10 minutes at 10,000 rpm. Samples of each gingival fluid will be analyzed for IL-1β, IL-4, IL-6, IL-8, IL-10, IL-17, TNFα and IFN-Δ by Luminex/MAGpix technology, which will not only determine the presence, but will quantify in absolute terms the concentration of different markers in the same sample, using commercially available kits, following the manufacturer's instructions. Briefly, samples will be diluted in PBS buffer + 5% Tween, and vortexed for 30 seconds, prior to analysis. After gentle centrifugation, 25 µL of supernatant will be placed in 96-well plates together with the immunolabeled beads specific for each cytokine/protease. After incubation with the beads, secondary antibodies and substrate will be provided, and the plates will be read using the MAGpix platform. The concentration of each analyte will be expressed in pg/µL. Samples with quantification below the detection limit of the analysis will be recorded as "zero", and samples above the quantification limit of the standard curve will be recorded with a value equal to the highest value of the curve.
7. Statistical Analysis: - Statistical analyses will be performed to compare clinical parameters, microbiome composition and cytokine expression between groups throughout the follow-up period. - The difference in efficacy between the two procedures will be assessed.

All analyses of this research will be performed in the research laboratories of the Periodontics area of the Piracicaba School of Dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are adult patients (over 18 years old), diagnosed with Peri-implantitis.

Exclusion Criteria:

* The following conditions will also be excluded: Pregnancy or lactation; Use of antibiotic or anti-inflammatory medication in the 6 months prior to the study; Presence of systemic diseases that make the surgical procedure impossible; Periodontal treatment including subgingival instrumentation in the 6 weeks prior to the study; Chronic alcohol users; Previous periodontal surgeries in the region of interest; Oral pathologies in the region of interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical parameters before and after implantoplasty and compare them to surgical access without implantoplasty. | Baseline; 1,3 and 6 months after procedure.
  Plaque index.
Clinical parameters before and after implantoplasty and compare them to surgical access without implantoplasty. | Baseline; 1,3 and 6 months after procedure.
  Bleeding on probing.
Clinical parameters before and after implantoplasty and compare them to surgical access without implantoplasty. | Baseline; 1,3 and 6 months after procedure.
  Probing depth.
Clinical parameters before and after implantoplasty and compare them to surgical access without implantoplasty. | Baseline; 1,3 and 6 months after procedure.
  Clinical insertion level.
Quantity of titanium particles in the crevicular fluid before and after implantoplasty. | Baseline; 1,3 and 6 months after procedure.
  Concentration of Titanium in the peri-implant environment.
To characterize and compare the peri-implant microbiological profile before and after implantoplasty. | Baseline; 1,3 and 6 months after procedure.
  Microbiome.

SECONDARY OUTCOMES:
Correlation between the presence of titanium particles, microbiological profile and local inflammatory response. | Baseline; 1,3 and 6 months after procedure.
  Evaluation and correlation of the results found in the clinical (clinical signs), microbiological (taxonomy of the species involved) and immunological evaluation (inflammatory cells most present) to better define the prognosis of each treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Renato Casarin, PhD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Piracicaba Dental School, Piracicaba, São Paulo, Brazil